CLINICAL TRIAL: NCT03087097
Title: Transfer of Healthy Gut Flora for Restoration of Intestinal Microbiota Via Enema (THRIVE) for Patients in the Rehabilitative Phase of Malnutrition: A Pilot Study Evaluating Microbial Engraftment, Safety and Nutritional Outcomes
Brief Title: Transfer of Healthy Gut Flora for Restoration of Intestinal Microbiota Via Enema for Patients in the Rehabilitative Phase of Malnutrition
Acronym: THRIVE
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: COVID-19 pandemic and resource constraints
Sponsor: Microbiome Health Research Institute (Other)
Collaborators: University of Cape Town (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: THRIVE001
Record Dates: First submitted 2016-12-12; First posted 2017-03-22 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Severe Acute Malnutrition; Moderate Acute Malnutrition
Keywords: SAM; MAM
MeSH Terms: conditions — Severe Acute Malnutrition | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Fecal Microbiota Transplant (Experimental): FMT by enema: 10mL/kg (maximum 150mL) of healthy donor human intestinal microbiota will be infused.
  Interventions: Biological: Fecal Microbiota Transplantation
- Standard of Care (No Intervention): Standard of care treatment for malnutrition as prescribed by local and national Department of Health Guidelines

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — Fecal microbiota delivered by rectal catheter enema in participants 12-60 months of age with malnutrition (MAM or SAM) who are in the rehabilitation phase of treatment and have failed to respond to at least 4 weeks of standard therapy.
  Other Names: Microbiota transfer therapy (MTT)
  Arms: Fecal Microbiota Transplant

SUMMARY:
This single-center, randomized, open-label trial will compare the safety of MTT delivered by rectal catheter enema in participants 12-60 months of age with malnutrition (moderate acute malnutrition [MAM] or severe acute malnutrition [SAM]) who are in the rehabilitative phase of treatment and have failed to respond to at least 4 weeks of standard therapy. Participants must meet inclusion criteria, no exclusion criteria prior to randomization. Participants will then be randomized in a 1:1 ratio at each site to 1 of 2 treatment groups:

* MTT by rectal catheter enema: 10mL/kg (maximum 150mL, +/- 5ml) of healthy donor human intestinal microbiota will be infused.
* Standard of care treatment for malnutrition as prescribed by local and national Department of Health Guidelines Participants will be evaluated through 56 days (±3) after randomization for primary outcomes (safety) as well as secondary outcomes (nutritional, clinical and microbiological response).

Participant blood and urine samples will be collected at enrollment and day 56. Participant stool samples will be collected at enrollment and through days 3, 7, 21 and 56, thereafter, 3 months, 4 months, and 6 months. A caregiver stool sample will be collected at enrollment and day 56. Samples will be used for microbiome determination and other exploratory microbiological endpoints. An aliquot of donor stool will also be stored for microbiome determination and other exploratory microbiological endpoints and assessment of newly acquired infectious agents.

ELIGIBILITY:
Participant Inclusion Criteria

Participants eligible to participate in this study must meet the following inclusion criteria:

1. Age 12 to 60 months.
2. Current diagnosis of malnutrition (defined as a WHZ less than -2 according to the WHO 2006 standards or a MUAC less than 125mm) with failure to respond nutritionally, defined as:

   a. A WHZ of less than -2 according or a mid-upper-arm circumference of less than 125 mm i. No medical complications present ii. Participant is sufficiently alert and successfully passes the appetite test which involves consumption of breastmilk or a ready to use therapeutic food (RUTF) under supervision.

   iii. Participant is in the rehabilitation phase of treatment for malnutrition
3. HIV negative
4. Received at last four weeks of optimal WHO treatment for malnutrition:

   1. Micronutrient supplementation (Vitamin A, zinc and iron) as recommended by local guidelines
   2. Nutritional rehabilitation as recommended by local guidelines.
5. Written informed consent obtained by parent or caregiver.

Participant Exclusion Criteria

Participants will not be able to participate if they meet any of the following exclusion criteria:

1. Evidence of current complicated malnutrition defined as any of the following:

   1. Admitted to acute care ward as inpatient
   2. Signs of severe acute infection such as pneumonia, bacteremia, meningitis. Minor infections such as candida dermatitis, pharyngitis, upper respiratory tract infections will be eligible for inclusion at the discretion of the study physician.
   3. One or more WHO Integrated Management of Childhood Illness danger signs.(3)
   4. Failure to pass appetite test.
   5. Presence of known comorbid diseases such as pulmonary Tuberculosis on treatment, cystic fibrosis, type I diabetes mellitus, intestinal malabsorptive syndromes, chronic lung disease, chronic liver disease, chronic renal disease, chronic neurological diseases (e.g. cerebral palsy) or malignancy undergoing active chemotherapy.
   6. Bilateral pitting pedal edema or generalized anasarca
2. Have taken antibiotics in the past seven days before the Day 0 visit or are anticipated to need antibiotics up to seven days before the Day 0 visit.
3. Congenital malformations, syndromic conditions, and congenital metabolic abnormalities (inborn errors of metabolism) that may adversely affect growth and in the view of the clinician, exposes the child to increased risk.

   a. Fetal alcohol syndrome (FAS) is not an exclusion.
4. Presence of bilateral pitting edema Grade 2.
5. Contraindications to rectal catheter enema:

   1. Anorectal malformations
   2. Rectal prolapse
   3. Hirschsprungs disease
   4. Other contraindication to enema.
6. Primary immune deficiencies
7. Acute, persistent or chronic diarrhea.
8. Dysentery
9. Intestinal abnormalities including malformations, Hirschsprungs disease and short bowel syndrome
10. Any condition that the physician investigators deems unsafe, including other conditions or medications that the investigator determines puts the participant at greater risk from MTT

Ages: 12 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 5 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Events | 56 days
  Number of participants with an Adverse Event grade 2 or above up to 56 days post-treatment

SECONDARY OUTCOMES:
Nutritional recovery: | 56 days
  Proportion of participants with nutritional recovery at day 56 after randomization. Defined as weight for height z-score (WHZ) ≥ -2 or MUAC ≥ 125 mm. In cases where there is a significant discrepancy between the weight and MUAC the participants weight will be used as the definitive measure.
Clinical: | 56 days
  Presence of signs and symptoms or complications of acute malnutrition. Clinical signs include fever (axillary temperature > 38.5⁰C), tachypnea (average of two measures; defined as respiratory rate of > 40 breaths per minute for children 12-60 months of age). Symptoms include diarrhea (≥ 3 loose stools in the last 24 hours), vomiting, and cough.
Microbiological: | 56 Days
  Assess engraftment of donor microbial communities in recipients through taxonomic characterization of donor and recipient microbiota pre- and post-MTT using both 16S rRNA and metagenomic techniques.
Translational: | 56 Days
  Assess the capacity for MTT to normalize biomarkers correlated with disease status and mortality in malnutrition. Stool biomarkers include Myeloperoxidase, Alpha-1-Antitrypsin, fecal calprotectin and neopterin. Serological biomarkers include CRP, endotoxin assay (Hek-Blue), and leptin.

CONTACTS AND LOCATIONS:
Overall Officials: Majdi A Osman, MD MPH, Principal Investigator — Microbiome Health Research Institute; Shrish Budree, MD MBChB DCH FCPeds, Principal Investigator — Microbiome Health Research Institute
Locations (1):
- University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Undecided